CLINICAL TRIAL: NCT00357656
Title: Antihemophilic Factor (Recombinant) Plasma/Albumin-Free Method (rAHF PFM): A Phase 3/4, Prospective, Controlled, Randomized, Multi-Center Study to Compare the Efficacy and Safety of Continuous Infusion (CI) Versus Intermittent Bolus Infusion (BI) in Subjects With Severe or Moderately Severe Hemophilia A Undergoing Major Orthopedic Surgery
Brief Title: Phase 3/4 Study of a Recombinant Protein-Free Factor VIII (rAHF-PFM): Comparison of Continuous Infusion Versus Intermittent Bolus Infusion in Hemophilia A Subjects Undergoing Major Orthopedic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Baxalta Innovations GmbH, now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 060402; 2005-005697-71 (EudraCT Number)
Record Dates: First submitted 2006-07-25; First posted 2006-07-27 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia A
Keywords: Hemophilia A (severe or moderately severe)
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BI (Experimental): Bolus infusion of rAHF-PFM
  Interventions: Drug: Recombinant Protein-Free Factor VIII (rAHF-PFM)
- CI (Experimental): Continuous infusion of rAHF-PFM
  Interventions: Drug: Recombinant Protein-Free Factor VIII (rAHF-PFM)

INTERVENTIONS:
Drug: Recombinant Protein-Free Factor VIII (rAHF-PFM) — An initial loading dose will be administered intravenously over a period <= 5 minutes (maximum of infusion rate of 10 mL/minute) within 60 minutes prior to surgery dose in order to maintain a minimum target FVIII level of at least 80% of normal.
  CI will start prior to surgery as soon as the loading dose has been administered, at a rate calculated according to a formula provided by the sponsor.
  All study product must be administered with a syringe pump running at an infusion rate according to the dosing regimen, but always >= 0.4 mL/h.
  Arms: CI
Drug: Recombinant Protein-Free Factor VIII (rAHF-PFM) — The treatment schedule for intermittent BI of rAHF-PFM will begin with the administration of the loading dose according to the dose recommendations provided by the sponsor. If required by the hemostatic challenge, additional boluses may be administered after a blood sample for FVIII determination has been drawn. All infusions of rAHF PFM will be given over a period <= 5 minutes (maximum infusion rate, 10 mL/min).
  Arms: BI

SUMMARY:
The purpose of this study is to compare the hemostatic efficacy and safety of continuous infusion versus intermittent bolus infusion in the peri- and post-operative setting, employing rAHF-PFM, a recombinant antihemophilic factor manufactured without added human or animal proteins, in previously treated patients with severe or moderately severe hemophilia A (baseline factor VIII level <= 2% of normal) who are undergoing unilateral major orthopedic surgery that requires drain placement. The total study period per subject (from consent to study completion) will vary from approximately 9 to 26 weeks and will involve clinical and laboratory assessments.

ELIGIBILITY:
Inclusion Criteria:

* The subject or the subject's legally authorized representative has provided signed informed consent.
* The subject is within 18 to 70 years of age.
* The subject has severe or moderately severe hemophilia A, defined by a baseline factor VIII level <= 2% of normal, as tested at screening. A subset of 15 subjects per group must have baseline factor VIII levels < 1% of normal.
* The aPTT must be within the range of normal after administration of FVIII concentrate, as determined in the preoperative pharmacokinetic evaluation, or as documented in the medical history, if available.
* The subject is scheduled to undergo an elective unilateral major orthopedic surgery that requires drain placement.
* The subject was previously treated with factor VIII concentrate(s) for a minimum of at least 150 exposure days (as estimated by the investigator) prior to study entry.
* Human immunodeficiency virus (HIV) positive subjects must be immunocompetent as determined with a CD4 count >= 200 cells/mm³ (CD4 count at screening), but HIV negative subjects with a CD4 count < 200 cells/mm³ qualify, if immunocompetency is documented.
* The subject has a life expectancy of at least 28 days from the day of surgery.

Exclusion Criteria:

* The subject has a detectable factor VIII inhibitor at screening, with a titer >= 0.4 BU (Nijmegen modification of the Bethesda assay) in the central laboratory.
* The subject has a history of factor VIII inhibitors with a titer >= 0.4 BU (by Nijmegen assay) or >= 0.5 BU (by Bethesda assay) at any time prior to screening.
* The subject is scheduled to undergo any other concurrent minor or major surgery during the course of the study. The placement of central venous lines and the performance of fine needle aspiration biopsies are permitted.
* Excluding hemophilia-related physical impairments, the subject is assigned to NYHA class >= III according to the New York Heart Association (NYHA).
* The subject has an abnormal renal function (serum creatinine > 1.5 mg/dL).
* The subject has active hepatic disease (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] levels > 5 times the upper limit of normal).
* The subject has severe chronic liver disease as evidenced by, but not limited to, any of the following: International Normalized Ratio (INR) > 1.4, hypoalbuminemia, portal vein hypertension including presence of otherwise unexplained splenomegaly and history of esophageal varices.
* The subject has clinical and/or laboratory evidence of abnormal hemostasis from causes other than hemophilia A (e.g., late-stage chronic liver disease, immune thrombocytopenia purpura).
* The subject is currently receiving, or is scheduled to receive during the course of the study, an immunomodulating drug other than anti-retroviral chemotherapy (e.g., alpha-interferon, corticosteroid agents at a dose equivalent to hydrocortisone greater than 10 mg/day).
* The subject has a known hypersensitivity to mouse or hamster proteins.
* The subject has received another investigational drug study within 30 days prior to screening and/or is scheduled to receive additional investigational drug during the course of the trial in the context of another investigational study.
* The subject is identified by the investigator as being unable or unwilling to cooperate with study procedures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2006-05-29 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2015-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (36):
- United States (10):
  - Los Angeles Orthopaedic Hospital, Los Angeles, California
  - Georgetown University, Washington D.C., District of Columbia
  - Rush Presbyterian St. Lukes, Chicago, Illinois
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Tulane University, New Orleans, Louisiana
  - Johns Hopkins Medical Institutions, Baltimore, Maryland
  - Brigham and Women´s Hospital, Boston, Massachusetts
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - The University of Texas Health Science Center at Houston Medical School, Houston, Texas
- University Hospital for Internal Medicine I (Hematology/Hemostaseology), Vienna, Austria
- Belgium (2):
  - Cliniques Universitaires St. Luc, Haematology Department, Brussels
  - University Hospital Gasthuisberg, Leuven
- Hôpital Edouard Herriot, Lyon, France
- Hungary (3):
  - State Health Centre, National Hemophilia Centre, Budapest
  - University of Debrecen, 2nd Dept of Internal Medicine, Debrecen
  - PTE ÁOK I. Internal Medical Clinic, Dept of Hematology, Pécs
- Italy (2):
  - Centro Emofilia e Trombosi "Angelo Bianchi Bonomi", Milan
  - Department of Clinical & Experimental Medecine, AOU Federico II, Naples
- Netherlands (3):
  - AMC Medical Research BV, Department of Vascular Medicine, Amsterdam
  - University Medical Centre Groningen, Groningen
  - Academic Hospital Maastricht, Maastricht
- Rikshospitalet, Oslo, Norway
- Poland (2):
  - Krakowskie Centrum Rehabilitacji, Krakow
  - Instytut Hematologii i Transfuzjologii, Klinika Zaburzeń Hemostazy i Chorób Wewnętrznych, Warsaw
- Portugal (2):
  - Centro Hospitalar de Coimbra, Coimbra
  - Hospital Santo António, Porto
- Romania (3):
  - Fundeni Clinical Institute, Clinical Laboratory "St. Berceanu" Hematology and Bone Marrow Transplantation Department, Bucharest
  - National Blood Transfusion Institute, Bucharest
  - "Louis Turcanu" Emergency Clinical Children´s Hospital, 3rd Pediatrics Department, Hemophilia Center, Timișoara
- Russia (3):
  - Regional Hemophilia Center, Kirov
  - Hematology Research Center under Russian Academy of Medical Sciences, Department of Reconstructive Orthopedic Surgery for Hemophilia Patients, Moscow
  - Russian Research Institute of Hematology and Transfusiology, Department of Surgical Hematology and Angiology, Saint Petersburg
- Spain (2):
  - Hospital Vall d´Hebron, Servei d´Hemofilia, Barcelona
  - Hospital Universitario La Fe, Valencia
- University Hospital MAS, Department for Coagulation Disorders, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conducted at 22 clinical sites in 12 countries (US, Austria, Norway, France, Portugal, Netherlands, Spain, Russia, Romania, Hungary, Italy, Poland). Of 85 participants enrolled, 72 participants participated in a PK study in the preoperative period; 63 participants were then randomized to treatment by continuous or bolus infusion.
Pre-assignment Details: Of 85 participants enrolled,15 were screen failures (2 after PK), 4 discontinued on the basis of the PK study in the preoperative period, 1 died, 1 was discontinued by physician decision (imprisonment), and 1 was discontinued per sponsor decision. Eventually, 63 participants were randomized to treatment by continuous (n=32) or bolus infusion (n=31)
Groups:
- Bolus Infusion: Bolus infusion of ADVATE (rAHF-PFM)
- Continuous Infusion: Continuous infusion of ADVATE (rAHF-PFM)
Period: Overall Study
Arm/Group | Bolus Infusion | Continuous Infusion
Started | 31 | 32
Completed | 31 | 29
Not Completed | 0 | 3
Not completed — Other, No surgery performed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bolus Infusion | Continuous Infusion | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 32 | 63
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.6 (9.76) | 39.0 (11.52) | 38.8 (10.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 31 | 32 | 63

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Packed Red Blood Cell (PRBC) Volume in the Drainage Fluid During the First 24 Hours Following Surgery in Subjects Receiving ADVATE (rAHF-PFM) by Bolus (BI) or Continuous Infusion (CI)
Description: Drainage fluid volume was to be measured cumulatively and recorded every 8 hours ± 30 minutes during the first 24 hours following surgery. Unit of measure: Tera per Liter is the PRBC concentration in 10^12 units per 1 liter of drainage fluid.
Time Frame: During the first postoperative 24 hours every 8 hours ± 30 minutes the drainage fluid was to be recorded..
Population: All subjects who were randomized to receive BI or CI and have observed drainage volumes up to 24 hours including hematocrit results for these drainage fluids. The overall number of participants treated by BI and CI comprises the number of participants in Stratum A, B and C for BI and CI.
Measure: Mean (Standard Deviation); unit: Tera per Liter
Groups:
- BI Stratum A: Participants who underwent unilateral knee replacement and were treated by bolus infusion
- BI Stratum B: Participants who underwent hip surgery and were treated by bolus infusion
- BI Stratum C: Participants who underwent shoulder/elbow/ankle/knee (except knee replacement) surgery and were treated by bolus infusion
- CI Stratum A: Participants who underwent unilateral knee replacement and were treated by continuous infusion
- CI Stratum B: Participants who underwent hip surgery and were treated by continuous infusion
- CI Stratum C: Participants who underwent shoulder/elbow/ankle/knee (except knee replacement) surgery and were treated by continuous infusion
Arm/Group | Bolus Infusion | Continuous Infusion | BI Stratum A | BI Stratum B | BI Stratum C | CI Stratum A | CI Stratum B | CI Stratum C
Number analyzed (Participants) | 28 | 26 | 22 | 2 | 4 | 23 | 1 | 2
Tera per Liter | 3.632 (0.971) | 3.383 (0.632) | 3.718 (0.978) | 2.855 (1.732) | 3.548 (0.577) | 3.345 (0.616) | 3.400 (NA) — Stratum B for continuous infusion has only one subject with available data, therefore standard deviation is not available. | 3.820 (1.103)
Statistical Analysis 1: Comparison: Bolus Infusion vs Continuous Infusion vs BI Stratum A vs BI Stratum B vs BI Stratum C vs CI Stratum A vs CI Stratum B vs CI Stratum C; The main analysis used a point estimate and a two-sided 95% confidence interval for ratio of the primary outcome measure of CI over BI combined over the three strata: stratum A: unilateral knee replacement, stratum B: hip surgery, stratum C: shoulder/elbow/ankle/knee (except knee replacement) surgery; Test type: Non-Inferiority or Equivalence — Non-inferiority by the 200% margin of non-inferiority was demonstrated if the upper confidence limit of a 95% 2-sided confidence interval for the ratio of means did not exceed 200%; p = 0.001, Hypothesis test — one-sided p-value against the null hypothesis of ration >=200%; Mean ratio CI/BI = 0.924, 95% CI 2-sided [0.816 to 1.046]

2. Secondary Outcome: Actual Postoperative Blood Loss During the First 24 Hours Compared With the Average Blood Loss as Predicted Preoperatively by the Operating Surgeon
Description: Drainage fluid volume was to be measured cumulatively and recorded every 8 hours ± 30 minutes during the first 24 hours following surgery. Prior to surgery, the operating surgeon was to predict the estimated duration of surgery and the volume (mL) of the estimated expected blood loss for the surgery in a hemostatically normal individual of the same sex, age, and stature as the study subject 1) for the intraoperative procedure (defined as the time period from incision to application of compressive dressing and release of tourniquet, if applicable), 2) for the first 24 hours postoperatively, and 3) for the postoperative period until drain removal, if drainage continued beyond 24 hours. Units: Milliliter of blood
Time Frame: During the first 24 postoperative hours blood loss was measured every 8 hours ± 30 minutes
Population: All subjects who were randomized to receive BI or CI and have observed drainage volumes up to 24 hours. The overall number of participants treated by BI and CI comprises the number of participants in Stratum A, B and C for BI and CI.
Measure: Mean (Standard Deviation); unit: Milliliter
Groups:
- Contiuous Infusion: Continuous infusion of ADVATE (rAHF-PFM)
Arm/Group | Bolus Infusion | Contiuous Infusion | BI Stratum A | BI Stratum B | BI Stratum C | CI Stratum A | CI Stratum B | CI Stratum C
Number analyzed (Participants) | 31 | 29 | 24 | 2 | 5 | 24 | 2 | 3
Milliliter | 709.28 (150.103) | 811.11 (79.511) | 724.48 (66.367) | 265 (49.497) | 814.03 (171.019) | 819.22 (66.992) | 713.49 (0) | 811.25 (163.027)

3. Secondary Outcome: Actual Postoperative Blood Loss Compared to the Expected Average Blood Loss Until Drain Removal as Predicted Preoperatively by the Surgeon
Description: The total blood loss for the postoperative period (from end of surgery until drain removal) was adjusted for the expected blood loss by applying a log-transformation of the blood loss data. The drainage volume was measured every 8 hours +/- 30 minutes during the first 24 hours. If the drainage continued beyond 24 hours, the PRBC volume and hemoglobin was to be measured cumulatively every 24 hours or whenever the drainage bottle was emptied and at the time of drain removal. Prior to surgery, the operating surgeon was to predict the estimated duration of surgery and the volume (mL) of the estimated expected blood loss for the surgery in a hemostatically normal individual of the same sex, age, and stature as the study subject for the first 24 hours postoperatively, and for the postoperative period until drain removal, if drainage continued beyond 24 hours. Units: Milliliter of blood
Time Frame: From end of surgery (application of compressive dressing and release of tourniquet, if applicable) until drain removal (up to postoperative day 7).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Bolus Infusion | Continuous Infusion | BI Stratum A | BI Stratum B | BI Stratum C | CI Stratum A | CI Stratum B | CI Stratum C
Number analyzed (Participants) | 30 | 28 | 23 | 2 | 5 | 23 | 2 | 3
Milliliter | 766.73 (182.463) | 929.49 (167.662) | 752.91 (42.343) | 341.5 (135.075) | 1000.37 (259.239) | 899.83 (45.459) | 921.1 (42.906) | 1162.48 (514.033)

4. Secondary Outcome: Number of Bleeding Episodes During Treatment With Continuous or Bolus Infusion
Description: To simplify the results below: Bleeding episodes were reported for 4 subjects (3 subjects on bolus infusion: 2 in Stratum A and 1 in Stratum B, and 1 subject on continuous infusion/Stratum B). The 4 subjects had 1 bleeding episode each. No bleeding episodes were reported for Stratum C.
Time Frame: Through Postoperative Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Bleeding Episodes
Groups:
- Bolus Infusion: Bolus infusion of rAHF-PFM
- Continuous Infusion: Continuous infusion of rAHF-PFM
Arm/Group | Bolus Infusion | Continuous Infusion | BI Stratum A | BI Stratum B | BI Stratum C | CI Stratum A | CI Stratum B | CI Stratum C
Number analyzed (Participants) | 31 | 29 | 24 | 2 | 5 | 24 | 2 | 3
Bleeding Episodes | 0.10 (0.301) | 0.03 (0.186) | 0.08 (0.282) | 0.50 (0.707) | 0.00 (0.000) | 0.00 (0.000) | 0.50 (0.707) | 0.00 (0.000)

5. Secondary Outcome: Number of Units of Packed Red Blood Cells Transfused
Time Frame: During the first postoperative 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: PRBC Units
Arm/Group | Bolus Infusion | Continuous Infusion | BI Stratum A | BI Stratum B | BI Stratum C | CI Stratum A | CI Stratum B | CI Stratum C
Number analyzed (Participants) | 31 | 29 | 24 | 2 | 5 | 24 | 2 | 3
PRBC Units | 0.9 (1.2) | 1.3 (1.4) | 1.0 (1.3) | 1.5 (2.1) | 0.2 (0.4) | 1.2 (1.3) | 3.5 (2.1) | 0.7 (1.2)

6. Secondary Outcome: Number of Adverse Events Related to the Administration of the Study Product.
Description: All AEs from the first study drug exposure until the study completion/discontinuation date were to be recorded. Each AE was to be evaluated by the investigator for causal relationship (i.e., unrelated, possibly related or probably related) to the study product.
Time Frame: From first study drug exposure until study completion/discontinuation (approximately 9-26 weeks per subject)
Population: Participants in the Safety Analysis Set treated with at least one ADVATE infusion.
Measure: Number; unit: Adverse Events
Groups:
- Safety Analysis Set: All participants treated with at least one ADVATE (rAHF-PFM) dose.
Arm/Group | Bolus Infusion | Continuous Infusion | Safety Analysis Set
Number analyzed (Participants) | 31 | 32 | 72
Adverse Events | 6 | 8 | 14

7. Secondary Outcome: Incidence of Factor VIII Inhibitory Antibody (≥0.4 Bethesda Units Using the Nijmegen Modification of the Bethesda Assay Formation)
Description: Number of participants that developed Factor VIII inhibitory antibody during the study.
Time Frame: Throughout the study period of approximately 9-26 weeks per participant
Population: Participants in the Safety Analysis Set treated with at least one ADVATE infusion.
Measure: Number; unit: Participants
Arm/Group | Bolus Infusion | Continuous Infusion | Safety Analysis Set
Number analyzed (Participants) | 31 | 32 | 72
Participants | 2 | 2 | 4

ADVERSE EVENTS:
Time Frame: Throughout the study period. Overall: 9 years and 6 months. Per participant: 9-26 weeks.
Groups:
- Bolus Infusion: All participants who were randomized to receive bolus infusion (BI) of ADVATE (rAHF-PFM). At total of 31 participants were randomized and received at least one ADVATE (rAHF-PFM) dose.
- Continuous Infusion: All participants who were randomized to receive continuous infusion (CI) of ADVATE (rAHF-PFM). At total of 32 participants were randomized and received at least one ADVATE (rAHF-PFM) dose.
- Not Assigned Participants: All participants who were not assigned to either bolus infusion or continuous infusion but received at least one ADVATE (rAHF-PFM) dose during pharmacokinetic evaluation. A total of 9 participants received only the pharmacokinetic infusion and were not randomized.
Arm/Group | Bolus Infusion | Continuous Infusion | Not Assigned Participants
Serious Adverse Events (participants affected / at risk) | 3/31 | 6/32 | 1/9
Other Adverse Events (participants affected / at risk) | 22/31 | 20/32 | 2/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bolus Infusion (N=31) | Continuous Infusion (N=32) | Not Assigned Participants (N=9)
Factor VIII inhibition (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle hemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bolus Infusion (N=31) | Continuous Infusion (N=32) | Not Assigned Participants (N=9)
Procedural pain (Injury, poisoning and procedural complications) | 10 (10) | 16 (16) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 10 (10) | 7 (7) | 1 (1)
Pyrexia (General disorders) | 10 (10) | 5 (5) | 0 (0)
Pain (General disorders) | 5 (5) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0)
Tooth Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle Hemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreements with PIs may vary per requirements of individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication. Baxalta requires a review of results communication (e.g. for confidential information) >= 30 days prior to submission. Baxalta may request an additional delay of <=120 days (e.g. for intellectual property protection).